CLINICAL TRIAL: NCT00596973
Title: Phase IV Study of Surgical Treatment of Type 2 Diabetes in Non-Morbidly Obese Patients
Brief Title: Surgical Treatment of Type 2 Diabetes in Non-Morbidly Obese Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AS07007
Record Dates: First submitted 2007-11-28; First posted 2008-01-17 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ileal transposition with SG (Experimental): Procedure: Surgical Treatment
  Interventions: Procedure: Surgical Treatment

INTERVENTIONS:
Procedure: Surgical Treatment — Ileal transposition with sleeve gastrectomy

SUMMARY:
The aim of this study is to assess the short term success and feasibility of ileal transposition with sleeve gastrectomy in non-morbidly obese patients with poorly controlled Type 2 Diabetes Mellitus

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed Type 2 Diabetes for 3 to 5 years.
2. Poorly controlled blood sugar despite standard of care* as demonstrated by HbA1c 8-11 for at least 6 months and 3 office visits. Standard of care is based on the ADA (American Diabetes Association) guidelines which include nutrition, exercise, education, behavior modification and pharmacological treatment. A co-investigator endocrinologist will ensure that the above standard of care has been met.
3. BMI between 25.0 and 34.4.
4. Stable weight as determined by no more than a 3% change in body weight in the last 3 months.
5. Age between 35 and 65 (both men and women will be included).
6. Able to provide Informed Consent.
7. Able to comply with follow-up procedures.

Exclusion Criteria:

1. Previous history of major abdominal surgery which may lead to a hostile abdomen.
2. Pregnancy
3. Patients who have an incurable malignant or debilitating disease
4. Serious uncorrectable impairment of coagulation (INR>1.4, PTT > + 3 secs), lungs, kidney or heart
5. Diagnosed severe eating disorder
6. Use of medication for weight loss in the last 6 months
7. Untreated endocrine disorder
8. Active peptic ulcer
9. Untreated H. pylori
10. Cognitive Impairment
11. Diabetic autonomic neuropathy
12. Symptomatic gastroparesis

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Treatment sucess based on patients' glycemic control | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Barry Salky, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States